CLINICAL TRIAL: NCT07353333
Title: Preliminary Evaluation of Clinical Application of SPECT Imaging Targeting GPC3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-250923
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: HCC; SPECT-CT

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sPECT imaging targeting GPC3 in malignant tumors (Experimental): Determine if targeting GPC3 SPECT is safe and effective method for imaging of malignant tumors.
  Interventions: Drug: 131I-aGPC3

INTERVENTIONS:
Drug: 131I-aGPC3 — Using targeted GPC3-specific imaging agents (e.g. , Iodine-131-aGPC3-Scfv) for integrated SPECTCT imaging, evaluate the pharmacokinetics distribution of the targeted drug in patients with hepatocellular carcinoma (HCC) by low-dose integrated diagnosis and treatment (i.e. , Iodine-131- imaging), and determine the metabolism, safety and tolerability of the drug in vivo

SUMMARY:
This project will target patients with highly clinically suspected or histopathology diagnosed hepatocellular carcinoma (HCC) using targeted GPC3-specific imaging agents (e.g. , Iodine-131-aGPC3-Scfv) for integrated SPECTCT imaging, to evaluate the pharmacokinetics distribution of the targeted drug in patients with hepatocellular carcinoma (HCC) by low-dose integrated diagnosis and treatment (i.e. , Iodine-131-RRB- imaging, to determine the metabolism, safety and tolerability of the drug in vivo Secondary objective: to evaluate the targeting of GPC3-SPECIFIC imaging agents in patients with hepatocellular carcinoma to assess the feasibility of this targeted agent for future treatment.

ELIGIBILITY:
Inclusion Criteria:

1. the subject or his/her legal representative can sign and date the informed consent form
2. commitment to follow the research procedures and cooperate in the implementation of the full-process research
3. patients with high clinical suspicion or histopathology diagnosis of HCC and generally in good condition
4. patients with a history of hepatocellular carcinoma who recur after treatment
5. women in their reproductive years were using contraception for at least one month before screening and were committed to using contraception throughout the study period and for the prescribed period after the end of the study

Exclusion Criteria:

1. inability to complete SPECTCT examination (including inability to lie down, claustrophobia, radiophobia, etc.)
2. acute systemic diseases and electrolyte disorders
3. patients with known hypersensitivity to GPC3 imaging agents or synthetic excipients
4. patients considered by the investigator to have poor adherence
5. pregnant or lactating patients
6. Have other factors not suitable to participate in this test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Radiation dose to human body | 1 year
  Metric/method of measurement：Use OLINDA/EXM software

SECONDARY OUTCOMES:
Region of Interest,ROI | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No